CLINICAL TRIAL: NCT01477775
Title: Customized Choice of P2Y12 Oral Receptor Blocker Based on Phenotype Assessment Via Point of Care Testing
Brief Title: Customized Choice of Oral P2Y12 Receptor Blocker
Acronym: PRU-MATRIX
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Italian Society of Invasive Cardiology (Other)
Collaborators: Eustrategy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFBU 13-I-PRU
Record Dates: First submitted 2011-10-27; First posted 2011-11-23 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Acute Coronary Syndrome; Coronary Angioplasty
Keywords: myocardial infarction; coronary stent; Oral P2Y12 receptor blocker; Platelet reactivity units (PRU)
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): The treating physician will be left free to give the oral P2Y12 receptor blocker, including clopidogrel,prasugrel or ticagrelor, which according to his/her clinical judgement is most appropriate for the individual patient.
  Interventions: Drug: Oral P2Y12 receptor blocker
- Customized choice of the oral P2Y12 receptor blocker (Experimental): The choice of the oral P2Y12 receptor blocker will be based on an algorithm which integrates phenotype information, including but not limited to residual on-treatment platelet reactivity assessed via Verifynow P2Y12 assay.
  Interventions: Drug: Customized choice for the oral P2Y12 receptor blocker

INTERVENTIONS:
Drug: Oral P2Y12 receptor blocker — Free choice among clopidogrel, prasugrel or ticagrelor
  Arms: Standard of Care
Drug: Customized choice for the oral P2Y12 receptor blocker — one drug among clopidogrel, prasugrel or ticagrelor based on an algorithm integrating phenotype information.
  Arms: Customized choice of the oral P2Y12 receptor blocker

SUMMARY:
A subset of patients recruited in the main MATRIX study will be randomized after intervention but before discharge to standard of care (the treating physician will decide which oral P2Y12 inhibitor will be added on top of aspirin) versus a customized approach based on an algorithm which integrates phenotypic information, including but not limited to residual on-treatment platelet reactivity assessed via VerifyNow P2Y12 Assay.

DETAILED DESCRIPTION:
Up to 20-30% of clopidogrel treated patients do not adequately respond to the drug and are at higher risk for ischemic events including death, myocardial infarction, stroke and stent thrombosis.

Residual high on-treatment platelet reactivity while the patient is on clopidogrel depends on a complex interplay of phenotypic (spontaneous platelet reactivity, inflammatory status, acuity of the clinical presentation, age, renal function) and genetic variables.

Two main Loss of function alleles have been identified: 1) CYP450 2C19*2 is present in around 25% of the Caucasian population and result in a lower amount of clopidogrel active metabolite. Carriers of 2C19*2 are at higher risk for death or MI and 2.7 fold increase in the risk of stent thrombosis if treated with conventional clopidogrel; 2) ABCB-1 C carriers have reduced clopidogrel absorption and they have similarly been shown to be at higher risk for ischemic adverse events if treated with clopidogrel. Many investigators have recently shown however, that the positive predictive value of genetic testing alone at the time of PCI is limited and the knowledge of genetic status alone with respect to the two previously described loss of function alleles is only poorly able to identify to long-term clopidogrel poor responders. An Algorithm has therefore been developed, combining phenotype information which has been shown to risk stratify both ischemic and bleeding events up to one year follow-up in PCI patients.

This algorithm has been developed from a single center retrospective registry. To prospectively validate it in the context of a prospective multicenter study, the first 320 patients recruited in the present study will undergo phenotype at discharge and at 30 days and genotype assessment at the time of randomization, irrespective of the group which they have been assigned to (i.e. standard of care or gene and phenotype). The hypothesis behind this mechanistic sub-study is that the use of this combined phenotype-genotype algorithm will increase the proportion of patients at 30 days who will be in the therapeutic range according to PRU values from 50% in the standard of care versus 70% in the gene and phenotype group.

ELIGIBILITY:
Inclusion Criteria:

* patients recruited in the main MATRIX study who underwent coronary angioplasty with stent placement.

Exclusion Criteria:

* unwillingness to sign this sub study specific informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death, myocardial infarction, stroke or BARC defined bleeding type 2, 3 or 5 | 1 year
  The time to first occurrence of any of the variables listed above will be reported as primary study outcome.
Proportion of patients in the therapeutic range for residual P2Y12 pathway activity according to PRU values. | 30 days
  We expect that the prospective use of the previously generated combined phenotype and genotype algorithm will result in an higher proportion of patients being in the therapeutic range with respect to the P2Y12 residual activity (70%) as compared to patients in who the P2Y12 inhibitor is left to the discretion of the treating physician. The first 320 patients recruited in the present study will participate into this mechanistic sub-study.

SECONDARY OUTCOMES:
Overall death | 1
cardiovascular death | 1 year
myocardial infarction | 1 year
stroke | 1 year
BARC bleeding type 2 | 1 year
BARC bleeding type 3 | 1 year
BARC bleeding type 5 | 1 year
Bleeding classified according to the Bleedscore | 1 year
Stent thrombosis | 1 year
  Stent thrombosis will be reported according to the ARC classification

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, MD, PhD, Principal Investigator — University Hospital of Ferrara
Locations (11):
- Italy (11):
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro, Calabria
  - University Hospital of Ferrara, Ferrara, Ferrara
  - Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan, MI
  - Spedali Civili di Brescia, Brescia
  - Azienda USL Sirai, Carbonia
  - Ospedale di Lodi, Lodi
  - Ospedale dei Colli, Cardiologia SUN, Naples
  - Ospedale degli Infermi di Rimini, Rimini
  - Ospedale San Giovanni Bosco, Torino
  - A. O. Ospedale Civile di Vimercate, Vimercate
  - Policlinico San Marco, Zingonia

REFERENCES:
- [Background] Campo G, Parrinello G, Ferraresi P, Lunghi B, Tebaldi M, Miccoli M, Marchesini J, Bernardi F, Ferrari R, Valgimigli M. Prospective evaluation of on-clopidogrel platelet reactivity over time in patients treated with percutaneous coronary intervention relationship with gene polymorphisms and clinical outcome. J Am Coll Cardiol. 2011 Jun 21;57(25):2474-83. doi: 10.1016/j.jacc.2010.12.047. PMID 21679849
- [Background] Campo G, Ferraresi P, Marchesini J, Bernardi F, Valgimigli M. Relationship between paraoxonase Q192R gene polymorphism and on-clopidogrel platelet reactivity over time in patients treated with percutaneous coronary intervention. J Thromb Haemost. 2011 Oct;9(10):2106-8. doi: 10.1111/j.1538-7836.2011.04457.x. No abstract available. PMID 21819538
- [Background] Campo G, Miccoli M, Tebaldi M, Marchesini J, Fileti L, Monti M, Valgimigli M, Ferrari R. Genetic determinants of on-clopidogrel high platelet reactivity. Platelets. 2011;22(6):399-407. doi: 10.3109/09537104.2011.579648. Epub 2011 May 31. PMID 21627411
- [Background] Valgimigli M, Campo G, de Cesare N, Meliga E, Vranckx P, Furgieri A, Angiolillo DJ, Sabate M, Hamon M, Repetto A, Colangelo S, Brugaletta S, Parrinello G, Percoco G, Ferrari R; Tailoring Treatment With Tirofiban in Patients Showing Resistance to Aspirin and/or Resistance to Clopidogrel (3T/2R) Investigators. Intensifying platelet inhibition with tirofiban in poor responders to aspirin, clopidogrel, or both agents undergoing elective coronary intervention: results from the double-blind, prospective, randomized Tailoring Treatment with Tirofiban in Patients Showing Resistance to Aspirin and/or Resistance to Clopidogrel study. Circulation. 2009 Jun 30;119(25):3215-22. doi: 10.1161/CIRCULATIONAHA.108.833236. Epub 2009 Jun 15. PMID 19528337